CLINICAL TRIAL: NCT03163914
Title: Comparison of the Effect of Epinephrine, Norepinephrine and Phenylephrine on Spinal Anesthesia Induced Hypotension
Brief Title: Effect of Vasopressors on Spinal Anaesthesia Induced Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Vasopressor
Record Dates: First submitted 2017-05-11; First posted 2017-05-23 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2017-11

CONDITIONS: Spinal Anesthesia
Keywords: vasopressor; spinal anaesthesia
MeSH Terms: interventions — Epinephrine; Norepinephrine; Phenylephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Partipicants and care providers will not known which medication will apply.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Epinephrine (Active Comparator): Epinephrine will prepare as 5µg/ ml and epinephrine infusion rate will adjust 30 ml/h.
  Interventions: Drug: Epinephrine
- Norepinephrine (Active Comparator): Norepinephrine will prepare as 5µg/ ml and epinephrine infusion rate will adjust 30 ml/h.
  Interventions: Drug: Norepinephrine
- Phenylephrine (Active Comparator): Phenylephrine will prepare as 100 µg/ ml and phenylephrine infusion rate will adjust 30 ml/h.
  Interventions: Drug: Phenylephrine
- Control (Placebo Comparator): Saline infusion will apply at equivalent volume till the surgical operation
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Epinephrine — Epinephrine infusion rate will adjust 30 ml/h (5µg/ ml )
  Other Names: group I
  Arms: Epinephrine
Drug: Norepinephrine — Norepinephrine infusion rate will adjust 30 ml/h (5µg/ ml )
  Other Names: group II
  Arms: Norepinephrine
Drug: Phenylephrine — Phenylephrine infusion rate will adjust 30 ml/h (100µg/ ml )
  Other Names: group III
  Arms: Phenylephrine
Drug: Saline — saline infusion will apply till the end of the surgery
  Other Names: group IV
  Arms: Control

SUMMARY:
160 pregnant patients will be enrolled in this study. Participants will divide in to 4 groups. Spinal anaesthesia will perform with 5% marcain heavy 2 ml+20 microgram fentanyl to the all patients. After performed spinal anaesthesia, vasopressor infusion will be started intravenously. Epinephrine will prepare 5 mg/ml and infusion rate will adjust 30 ml/h for Group E. Norepinephrine will prepare 5 mg/ml and infusion rate will adjust 30 ml/h for Group NE and 0.9% saline (group S) was launched immediately after induction of spinal anesthesia. Phenylephrine will prepare 100 microg/ml and infusion rate will adjust 30 ml/h for Group P. If systolic blood pressure decrease 20% of basal value or below to 100 mmHg, bolus ephedrine will apply intravenously (IV). If heart rate will decrease 60 beat per min or 20% of basal value, atropine will apply IV.

DETAILED DESCRIPTION:
After approved informed consent, 160 pregnant (term) patients with American society of anaesthesiologist (ASA) physiological status I-II will include this prospective, randomized clinical study. For randomisation of participants, computerized randomisation programme will use and they will divide into 4 groups. Basal value of systolic blood pressure(SBP) and heart rate (HR) will calculate with mean of the measure of 3 time SBP and HR before spinal anaesthesia. Spinal anaesthesia will perform with 5% marcain heavy 2 ml+20 microgram fentanyl at the point of lumbar 3-4 or 4-5 interspinous space to the all patients. After performed spinal anaesthesia, vasopressor infusion will start intravenously. Epinephrine, norepinephrine and phenylephrine will use for vasopressor infusion. Epinephrine will prepare 5 mg/ml and infusion rate will adjust 30 ml/h for Group E. Norepinephrine will prepare 5 mg/ml and infusion rate will adjust 30 ml/h for Group NE. Phenylephrine will prepare 100 microg/ml and infusion rate will adjust 30 ml/h for Group P. salin infusion will launch 30 ml/h for group Salin. If systolic blood pressure decrease 20% of basal value or below to 100 mmHg, bolus ephedrine will apply intravenously (IV) for rescue drug. If heart rate will decrease 60 beat per min or 20% of basal value, atropine will apply IV.

At the end of the study all collected data will use for statistically analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status
* Pregnant patients
* Full term pregnant

Exclusion Criteria:

* ASA III-IV physical status
* Emergency status
* Heart disease
* Hypertension
* Body mass index>25

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant patients
Enrollment: 160 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative maternal hypotension | At the time from start of vasopressor infusion till the end of surgery. The time frame is approximately 1 hour, peroperatively.
  The incidence of hypotension (described as less than 80% of baseline (prenatal) SBP or SBP <90 mm Hg), the total number of hypotension episodes during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hakkı Ünlügenç, Study Director — Cukurova University
Locations (1):
- Çukurova University Balcalı Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No